CLINICAL TRIAL: NCT02768064
Title: Temporary Pacemaker in Transcatheter Aortic Valve Implantation Patients
Acronym: PAMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Orlev Amir, Dr, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 065015-HMO-CTIL
Record Dates: First submitted 2016-02-10; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible screwed electrode (Experimental): In the TAVI patients, during the intervention procedure, a temporary pacemaker will be implanted, using a flexible screwed electrode.
  Interventions: Device: temporary pacemaker insertion
- Stiff standard electrode (Active Comparator): In the TAVI patients, during the intervention procedure, a temporary pacemaker will be implanted, using a stiff standard temporary electrode
  Interventions: Device: temporary pacemaker insertion

INTERVENTIONS:
Device: temporary pacemaker insertion — Insertion of pacemaker electrode (Medtronic flow direct pacing catheter), connect to external pacemaker (Medtronic).

SUMMARY:
During Transcatheter aortic valve implantation (TAVI) procedure, a new valve is implanted. The valve can be CoreValve (Medtronic Company) or Edward SAPIENS (Edwards Company).

All TAVI patients require a temporary pacemaker(PMK), which is usually performed by insertion of a standard temporary electrode through the femoral vein. The temporary PMK is associated with a small but significant rate of complications.

The PMK is usually removed immediately at the end of the TAVI procedure, only when using the Edward SAPIENS valve. The CoreValve valve is more associated with conduction complications, and thus the PMK is later removed in these cases.

PMK Complications seen include:

* Right Ventricle perforation by temporary electrode, leading to Pericardial bleeding, in some cases with Tamponade
* Infection
* Electrode dislocation causing In-effective pacing (and/or sensing)
* Prolonged bed rest
* Prolonged hospitalization
* Access related problems (hematoma, pneumothorax) In a review of a large cohort (1) of patients from Milan (JACC 2012) the rate of tamponade was 4.3% most of which was associated with the temporary PMK.

DETAILED DESCRIPTION:
The investigators had experienced not infrequent occurrences of temporary electrode associated tamponade, either acutely after Transcatheter aortic valve implantation (TAVI) completion, or delayed, in association with the electrode removal.

The tamponade rate in patients with a temporary pacemaker(PMK) was 14/150 (9.3%). Not all tamponade cases were related to the temporary PMK, 2 occurred in the setting of catastrophic annular rupture and one of the first cases was related to the Left Ventricle stiff wire.

The investigators also noted a significant prolongation of bed rest and hospital stay in patients with temporary PMK.

Using a flexible permanent pacing electrode which is actively fixed to the Right Ventricle and is placed through the jugular vein will reduce pacing-related complication rates (due to the flexibility of the electrode), time to ambulation (due to the fixation of the electrode), hospital stay and also unnecessary PMK. Cost will also be reduced due to prevention of complications and reduction in Intensive Cardiac Care Unit time.

Procedure time might be slightly prolonged since the placement of the standard electrode is more timely, however this prolongation is negligible, and the benefits of the flexible permanent pacing electrode are worth this prolongation

ELIGIBILITY:
Inclusion Criteria:

* All TAVI patients

Exclusion Criteria:

* Existing contraindication for either femoral or jugular venous access
* Refused informed consent
* Permanent PMK
* Platelets count less than 50 K.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pericardial effusion with or without tamponade | 1 week
  Pericardial effusion estimated by echocardiography, will be done during the hospitalization. It will be described as minimal/mild/moderate/large
Number of participants with Electrode Dislocation | 1 week
  Electrode Dislocation (sensing / pacing problems, requiring lead re-positioning).
  The dislocation will be diagnosed by chest X ray or by sensing / pacing parameters.
Number of participants with Bleeding complications | 1 week
  Bleeding complications, described as local hematoma within the area of the electrode insertion, during the procedure or the hospitalization.
Number of participants with Infections complications | 1 week
  Infections complications, described as fever above 38.0 celsius degree or positive blood culture during the hospitalization after the procedure.
Number of participants with access site complications | 1 week
  Access site complications describe as perforation of near organs (jugular artery)
Number of participants with Pneumothorax | 1 week
  Pneumothorax diagnosed by clinical examination and CXR within 3 days after the procedure.
Number of participants with pacemaker failure | 1 week
  Rates of Pacing or sensing failure during the procedure, or the days after,

SECONDARY OUTCOMES:
An implantation of permanent pacemaker | one year
  An implantation of permanent pacemaker (of any company, of any reason) within a year after TAVI in any hospital. The data will be collect from the hospital medical record system, and the patient report
The time (in days) the patient was able to get down from his bed to a chair, after the procedure | week
  The number of days from the TAVI procedure to the first time the patient was able to get down from his bad and sit on a chair. The data will be collected from the nurse description in the medical record.
The time (in days) the patients has stayed in Intensive Cardiac Care Unit | 2 weeks
  The number of days the patient was hospitalized in Intensive Cardiac Care Unit. The number will be calculated from the end of the TAVI procedure, till the patient went home or moved into the Cardiology department.
The Cost of Pacing equipment | 1 week
  Will be calculate by the sum of the electrode cost and the vascular shith cost
The TAVI procedure time | 1 day
  Will be taken from the technician report of starting and ending of the TAVI procedure
The TAVI fluoroscopic time | 1 day
  Will be taken from technician report of Fluoroscopic time
The permanent pacemaker activation (if implanted) | 1 year
  If a pacemaker was implanted to the patient, the data will be collected from the interrogation of the pacemaker.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Orlev, Dr, Principal Investigator — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webb JG, Wood DA. Current status of transcatheter aortic valve replacement. J Am Coll Cardiol. 2012 Aug 7;60(6):483-92. doi: 10.1016/j.jacc.2012.01.071. Epub 2012 Jun 27. PMID 22749306
- [Background] Barbash IM, Waksman R, Pichard AD. Prevention of right ventricular perforation due to temporary pacemaker lead during transcatheter aortic valve replacement. JACC Cardiovasc Interv. 2013 Apr;6(4):427. doi: 10.1016/j.jcin.2013.01.135. No abstract available. PMID 23597613
- [Background] Rezq A, Basavarajaiah S, Latib A, Takagi K, Hasegawa T, Figini F, Cioni M, Franco A, Montorfano M, Chieffo A, Maisano F, Corvaja N, Alfieri O, Colombo A. Incidence, management, and outcomes of cardiac tamponade during transcatheter aortic valve implantation: a single-center study. JACC Cardiovasc Interv. 2012 Dec;5(12):1264-72. doi: 10.1016/j.jcin.2012.08.012. PMID 23257375